CLINICAL TRIAL: NCT03599882
Title: Non-invasive Assessment of Liver Steatosis and Stiffness in HIV-infected Patients With Controlled Attenuation Parameter and Transient Elastography
Brief Title: Liver Steatosis and Stiffness in HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Cheng Chen, Associate professor, Chang Gung Memorial Hospital
Other Study IDs: HIV-LSM-CAP
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections; Fatty Liver; Liver Fibroses
Keywords: human immunodeficiency virus; liver steatosis; liver fibrosis; controlled attenuation parameter; transient elastography
MeSH Terms: conditions — HIV Infections; Fatty Liver; Liver Cirrhosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fibroscan — Fibroscan with controlled attenuation parameter and transient elastography

SUMMARY:
Background:

With the advances in treatment and clinical care, individuals with human immunodeficiency virus (HIV) infection have experienced an increase in life expectancy. Liver disease is common among HIV-infected patients due to the shared routes of transmission of HIV and viral hepatitis. Nonalcoholic fatty liver disease (NAFLD) is the most common cause of elevated aminotransferases in HIV-monoinfected adults without HBV or HCV.

Vibration-controlled transient elastography (VCTE) has been shown to have good sensitivity and specificity for assessment of liver fibrosis in HIV and viral hepatitis coinfected patients, as well as in HIV-negative NASH population. Controlled attenuation parameter (CAP), a novel physical parameter developed using the postulate that fat affects ultrasound propagation, measures the ultrasound attenuation at the center frequency of the FibroScan®.

Study design:

This is a prospective observational study.

Objective:

The aim of this study is to evaluate the liver steatosis and fibrosis in HIV-infected patients by noninvasive methods of VCTE and CAP.

Methods:

Patient number: 200

Inclusion criteria:

1. Age: 20-65 years
2. Males and females with HIV infection diagnosed by infection doctors
3. Willing and able to comply with the study requirements
4. Willing and able to provide written informed consent to participate in the study

Exclusion criteria:

1. Pregnancy
2. Unable to complete the noninvasive procedure of VCTE and CAP
3. Unwilling to provide written informed consent to participate in the study

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-65 years
2. Males and females with HIV infection diagnosed by infection doctors
3. Willing and able to comply with the study requirements
4. Willing and able to provide written informed consent to participate in the study

Exclusion Criteria:

1. Pregnancy
2. Unable to complete the noninvasive procedure of VCTE and CAP
3. Unwilling to provide written informed consent to participate in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV infection
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The changes of liver steatosis in HIV-infected patients by FibroScan (CAP) | 2 years
  The liver steatosis will be evaluated by controlled attenuation parameter at 6-month interval. The overtime changes will be explored.
The changes of liver fibrosis in HIV-infected patients by Fibroscan (VCTE) | 2 years
  The liver fibrosis will be assessed by transient elastography at 6-month interval. The overtime changes will be explored.

SECONDARY OUTCOMES:
The association between FIB-4 and liver fibrosis | 2 years
  FIB-4 will be calculated by a formula. FIB-4=[age(year)*AST(U/L)]/[platelet count*ALT(U/L)^0.5]
The association between BMI and liver steatosis | 2 years
  BMI is combination of BW and BH and presented as kg/m^2.
The association between lipid profile and liver steatosis | 2 years
  Lipid profile includes cholesterol, triglyceride, HDL cholesterol, LDL cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Cheng Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No